CLINICAL TRIAL: NCT05170373
Title: Effects of Ultrasound Guided Erector Spinae Plane Block in Radical Prostatectomy Surgery on Pain and Surgical Stress Response
Brief Title: ESP Block in Radical Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Damla Turan, Principal Investigator, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstanbulMU ESPB
Record Dates: First submitted 2021-11-03; First posted 2021-12-28 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Erector Spinae Plane Block
Keywords: Erektor Spinae Plane Block; Postoperative Analgesia; Surgical Stress Response

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP group (Active Comparator)
  Interventions: Procedure: ESP block
- control group (No Intervention)

INTERVENTIONS:
Procedure: ESP block — Before general anesthesia, ESP block was applied from the T12 vertebra level with 10 ml 0.5% bupivacaine HCL 5 ml 2% lidocaine HCL 5 ml 0.9% isotonic NaCl mixture
  Arms: ESP group

SUMMARY:
Our study aimed to examine the effects of ultrasound guided erector spinae plane block in radical prostatectomy surgery on pain and surgical stress response, to reduce adrenocortical and sympathetic discharge due to anesthesia and surgery, and to reduce peroperative opioid analgesic consumption.

DETAILED DESCRIPTION:
In this study 46 patients between the ages of 30-74, American Society of Anesthesiologists (ASA) score I-II and undergoing radical prostatectomy surgery at T.R. Ministry Of Health İstanbul Göztepe Prof. Dr. Süleyman Yalçın City Hospital were included. The patients were randomly divided into two groups as ESPB applied Group B (n=23) and not Group K (n=23). Patient-controlled analgesia (PCA) was initiated in all patients for postoperative analgesia. Patients' demographic data (age, gender, ASA score), intraoperative hemodynamic data, intraoperative and postoperative additional narcotic consumption, postoperative Numeric Rating Scale (NRS) scores (postoperative 0, 5 and 20 minutes and Then, 1, 3, 6, 12, 18 and 24 h), postoperative nausea-vomiting scores and possible complications related to block and / or surgery were recorded.Intraoperative MAP, HR, SpO2, BIS values of patients in both groups were recorded every 5 minutes. Blood glucose, insulin, cortisol, prolactin and C-reactive protein (CRP) were studied three times; preop morning at 6:00, intraoperative when surgical incision closing and postoperative 24h. in order to evaluate the surgical stress response in the patients.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II

Exclusion Criteria:

* diabetes
* coagulopathy
* local anesthetic
* drug allergy
* long hospitalization history,
* hormone disorder
* advanced organ failure
* history of steroid use
* vertebral anomalies
* mental retardation

Ages: 30 Years to 74 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Scale | postoperative 24 hours.
  Between 1-10. 1: no pain, 10: worst possible pain
Blood glucose | postoperative 24 hours.
  mg /dL
insulin | postoperative 24 hours.
  µIU/mL
cortisol | postoperative 24 hours.
  µg/dL
prolactin | postoperative 24 hours.
  µg/L
C-reactive protein | postoperative 24 hours.
  mg/L

SECONDARY OUTCOMES:
Remifentanil Consumption Speed | 3 hours
  µg /kg/dk

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Suleyman Yalcin City Hospital, Istanbul, Turkey (Türkiye)